CLINICAL TRIAL: NCT06944340
Title: Evaluating the Impact of World Health Organization Trauma Care Checklist on Clinical Outcome of Patients: A Prospective Randomized Controlled Trial
Brief Title: Evaluating the Impact of WHO Trauma Care Checklist on Clinical Outcome of Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Rao Erbaz Hassan, Trainee Medical Officer, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 526/DME/KMC
Record Dates: First submitted 2025-04-15; First posted 2025-04-25 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Trauma Related Injuries; Trauma
Keywords: Trauma; Trauma Outcomes; WHO Trauma Care Checklist; Trauma Checklist; Injury; Emergency Care
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Two-group, single-blinded, parallel assignment randomized controlled trial. Patients are randomly allocated to either receive standard trauma care (control group) or standard care enhanced with the WHO Trauma Care Checklist (intervention group). Outcomes are compared between groups over a 1-month follow-up period.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Trauma Care (No Intervention): Patients receive routine trauma care adhering to the hospital's existing protocols without using the WHO Trauma Care Checklist. Treatment includes stabilization, diagnostics, surgical/non-surgical interventions, and post-operative care as per institutional standards.
- WHO Trauma Care Checklist-Guided Care (Experimental): Patients receive trauma care guided by the WHO Trauma Care Checklist. The checklist is systematically applied by trained clinicians at critical stages of care (e.g., admission, pre-operative, post-operative, and discharge phases) to ensure adherence to evidence-based practices, including airway management, hemorrhage control, infection prevention, and monitoring for complications.
  Interventions: Other: WHO Trauma Care Checklist

INTERVENTIONS:
Other: WHO Trauma Care Checklist — A standardized checklist developed by the WHO for trauma care, designed to reduce errors and ensure compliance with critical steps in trauma management.
  Implemented by trained clinicians during patient assessment and treatment phases. Components include verification of patient identity, assessment of airway/breathing/circulation, pain management, monitoring for missed injuries, and post-resuscitation care. Checklist use is documented in medical records.
  Arms: WHO Trauma Care Checklist-Guided Care

SUMMARY:
This study is being conducted at the Department of Trauma and Orthopedics at Khyber Teaching Hospital, Peshawar. It will test whether using the World Health Organization (WHO) Trauma Care Checklist can help improve the care and recovery of patients who have experienced physical injuries (trauma).

Injuries are a major cause of death and disability, especially in countries like Pakistan. When someone is seriously injured, doctors must act quickly and carefully to save lives and prevent long-term problems. Checklists are simple tools that help healthcare providers make sure nothing is missed during treatment.

In this study, adult trauma patients will be randomly divided into two groups:

One group will receive the standard trauma care (Group A). The other group will receive trauma care with the help of the WHO checklist (Group B).

Doctors will compare the outcomes of both groups by looking at things like pain levels, injury severity, recovery progress, complications (like infections or organ problems), and overall satisfaction. The goal is to see if the checklist makes a meaningful difference in patient recovery and safety.

DETAILED DESCRIPTION:
Background

Trauma is one of the leading causes of mortality and long-term disability worldwide. In Pakistan, the burden of traumatic injuries is significant, especially among younger individuals. Contributing factors include road traffic accidents, workplace injuries, natural disasters, and violence. Despite being preventable and manageable in many cases, the lack of standardized emergency protocols and system-level interventions has resulted in suboptimal trauma care and increased complications. The WHO developed the TCC to support healthcare providers in delivering consistent, high-quality trauma care, especially in resource-limited settings.

Objective

This study aims to evaluate whether implementing the WHO Trauma Care Checklist during the initial assessment and management of trauma patients improves clinical outcomes compared to standard care alone. The primary hypothesis is that the checklist will help reduce complications, improve injury assessment accuracy, and enhance patient satisfaction.

Study Design and Setting

This is a prospective, single-blinded, randomized controlled trial being conducted at the Department of Trauma and Orthopedics, Khyber Teaching Hospital, Peshawar. The study will be conducted over six months following ethical approval.

Participants

A total of 60 adult trauma patients (aged 18-60 years) who meet specific inclusion criteria will be enrolled using simple random sampling. Participants will be randomly allocated to one of two groups:

Group A: Standard trauma care without the WHO checklist Group B: Standard trauma care with the WHO checklist Patients with severe comorbidities, pregnancy, chemotherapy, chronic mental illness, or substance abuse will be excluded.

Intervention

The WHO Trauma Care Checklist will be used by the clinical team during the initial management of patients in Group B. The checklist includes key safety steps related to airway, breathing, circulation, disability assessment, and exposure/environment, along with other evidence-based practices to prevent missed injuries and reduce medical errors.

Data Collection and Tools

Baseline demographic and clinical data will be collected at admission. Outcome assessments will include:

Improvement in Injury Severity Score (ISS) Visual Analogue Scale (VAS) for pain Glasgow Coma Scale (GCS) Duration of hospital stay and number of bed-bound days Occurrence of complications (e.g., sepsis, renal failure, pneumonia, wound infection) Mortality Missed injuries at presentation Patient satisfaction (rated on a 1-10 scale) Medical charts, direct observation, and patient interviews will serve as the primary data sources. Injury severity will be assessed by trained researchers using a standardized scoring system.

Follow-Up

Patients will be followed during their hospital stay and for one month post-discharge through phone calls or in-person visits. All outcomes will be assessed both at discharge and during the follow-up period.

Data Analysis

SPSS will be used for statistical analysis. Descriptive statistics will summarize patient characteristics and clinical outcomes. Independent t-tests and chi-square tests will compare outcomes between groups. A significance level of p < 0.05 will be used.

Significance

The results of this trial will help determine whether the WHO Trauma Care Checklist improves trauma care quality and outcomes in a low-resource hospital setting. If effective, the checklist could be implemented more widely to enhance trauma care across similar settings.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old
* Glasgow Coma Scale (GCC) equal to or more than 10
* Consenting to participate in the study

Exclusion Criteria:

* Patients who do not meet the inclusion criteria
* Patients who refrain from continuing the study
* Patients with the incomplete checklist
* Pregnancy
* History of chronic mental illness, lung or kidney disease
* Undergoing chemotherapy.
* Illicit drug dependency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-26 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Improvement in Injury Severity Score (ISS) | Assessed at admission and after initial management.
  difference in ISS at admission and after initial management. A higher difference means a better outcome.
Glasgow Coma Scale (GCS) Score | Measured at presentation and 1 hour post-treatment.
  Consciousness levels of participant. Average change/rise/fall. Higher GCS means better outcome
level of Pain | Assessed after initial management.
  Pain levels using the Visual Analogue Scale (VAS). A lower VAS score means better outcome.

SECONDARY OUTCOMES:
All-Cause Mortality Rate | 1 month post-treatment.
  Incidence of death within 1 month post-trauma.
Incidence of Post-Trauma Complications | 1 month post-treatment
  Rates of complications (e.g., cardiac arrest, pneumonia, pulmonary embolism, sepsis, wound infections).
Number of Bed-Bound Days | From admission to discharge (up to 1 month)
  Duration of immobilization during hospitalization
Patient Satisfaction Score | Assessed at 1 month follow-up.
  Patient-reported satisfaction with care quality on a scale of 1-10. Higher scores mean better outcomes.
Rate of Missed Injuries | Identified during 1-month follow-up.
  Proportion of injuries undetected during initial assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department, Khyber Teaching Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hyder AA, Razzak JA. The challenges of injuries and trauma in Pakistan: an opportunity for concerted action. Public Health. 2013 Aug;127(8):699-703. doi: 10.1016/j.puhe.2012.12.020. Epub 2013 Mar 13. PMID 23489711
- [Background] Bidhendi S, Ahmadi A, Fouladinejad M, Bazargan-Hejazi S. Evaluating implementation of WHO Trauma Care Checklist vs. modified WHO checklist in improving trauma patient clinical outcomes and satisfaction. J Inj Violence Res. 2021 Jan;13(1):5-12. doi: 10.5249/jivr.v13i1.1579. Epub 2020 Aug 16. PMID 32868497